CLINICAL TRIAL: NCT02280590
Title: Comparison of the Efficacy and Safety of Cresnon® and Crestor® in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNT_HLP_IV
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Rosuvastatin Calcium

ARMS (2):
- Cresnon® (Experimental): Rosuvastatin 10mg, tablet, q.d.
  Interventions: Drug: Rosuvastatin(Cresnon®)
- Crestor® (Active Comparator): Rosuvastatin 10mg, tablet, q.d.
  Interventions: Drug: Rosuvastatin(Crestor®)

INTERVENTIONS:
Drug: Rosuvastatin(Cresnon®) — 10mg
  Arms: Cresnon®
Drug: Rosuvastatin(Crestor®) — 10mg
  Arms: Crestor®

SUMMARY:
Comparison of the efficacy and safety of Cresnon® and Crestor® in patients with hyperlipidemia

- 8-week, active-controlled, open-label, randomized, parallelgroup, fixed-dose, noninferiority, multicenter, phase 4 design

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20
* Persons who have not reached LDL-C targeted level in accordance with the treatment guidelines for dyslipidemia released by Korean Society of Lipidology and Atherosclerosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The percent change in LDL-C | After taken medication for 8 weeks

SECONDARY OUTCOMES:
The percent change in total cholesterol, Triglyceride, HDL-C, non-HDL-C, and non-HDL-C/HDL-C | After taken medication for 8 weeks
The proportion of subjects reaching LDL-C targeted level in accordance with the treatment guidelines for dyslipidemia released by Korean Society of Lipidology and Atherosclerosis | After taken medication for 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea